CLINICAL TRIAL: NCT02740751
Title: Efficacy of Herbal Galactogogues on Weight Gain of the Newborns Within the First Month of Life in Breastfeeding Mothers
Brief Title: Efficacy of Herbal Galactogogues in Breastfeeding Mothers
Acronym: Galactogogue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, MD, Assoc Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SamiUlusCH-trials-stilltee
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Still-Tee (Active Comparator): Generic name: galactogoe herbal tee, still-tee Dosage: Three cups (each 200 ml) of tea of Still-Tee galactogogue tea will be used Frequency: Three times in a day Duration: for 4 weeks after birth
  Interventions: Dietary Supplement: Still-Tee
- Placebo (Placebo Comparator): The mothers of the babies will receive placebo tea which does not contain galactogogue herbs
  Interventions: Dietary Supplement: Still-Tee
- Water (No Intervention): The mothers of the babies will receive water

INTERVENTIONS:
Dietary Supplement: Still-Tee — The mothers of the babies will receive Still-Tee galactogogue tea
  Arms: Placebo; Still-Tee

SUMMARY:
Herbal teas with galactogoge effects have been used extensively in recent years in order to increase the amount of breast milk in lactating mothers. We also investigated whether a sleep-induced herbal tea (Still-Tee; Mamsel®) was effective in regulating the sleep of these mothers. Plain water was used as placebo.

DETAILED DESCRIPTION:
Herbal teas with galactogoge effects have been used extensively in recent years in order to increase the amount of breast milk in lactating mothers. Mothers of premature babies often have problems in breastfeeding and this study was designed to investigate if such herbal teas has any effect on the increasing of breast milk in mothers of premature babies. We also investigated whether a sleep-induced herbal tea (Still-Tee; Mamsel®) was effective in regulating the sleep of these mothers. Plain water was used as placebo.

ELIGIBILITY:
Inclusion Criteria:

* Babies with gestational age of 35-42 weeks
* Breasfed babies
* Lactating mothers
* Babies admitted to outpatient clinics of neonatology within the the first week of life

Exclusion Criteria:

* Babies with gestational age of <35 weeks
* Not breast feeding mothers
* Babies admitted to outpatient clinics of neonatology within the the first week of life

Ages: 3 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Weight gain | 4 weeks

SECONDARY OUTCOMES:
Breast milk volume | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, Assoc Prof, Study Director — Dr Sami Ulus Research and Training Hospital
Locations (1):
- Dr Sami Ulus Children Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208